CLINICAL TRIAL: NCT01437956
Title: Acute Bronchiolitis in Infants: Analysis of a Biomarker of Epithelial Lung Injury - Clinical and Virological Correlation
Brief Title: KL-6 Protein as a Biomarker of Lung Injury in Viral Bronchiolitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0104
Record Dates: First submitted 2011-09-12; First posted 2011-09-21 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Acute Viral Bronchiolitis
Keywords: Calcineurin; Bronchiolitis; Epithelial lung injury; Rhinovirus; Respiratory Syncytial Virus; Asthma
MeSH Terms: conditions — Bronchiolitis; Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Serum KL-6 protein has been described as a biomarker of epithelial lung injury in Respiratory Syncytial Virus bronchiolitis. The investigators can imagine that epithelial injury intensity has consequences on immediate and later respiratory prognosis. Furthermore, this prognosis seems to be different according to the respiratory causative virus. The investigators propose to study, during an epidemic season, the correlation between KL-6 levels and clinical severity, and the type of viral infection.

DETAILED DESCRIPTION:
Prospective, monocentric, case-control and transversal study Primary end-point: correlation between serum KL-6 level and severity of the bronchiolitis, evaluated by a clinical scoring system established at the time of the admission in Paediatric Emergency Unit Secondary end-points: respiratory virus detected by EIA and RT-PCR, phylogenetic study of rhinovirus, length of hospitalisation, immediate morbidity and mortality, risk of asthma at the age of three years old.

ELIGIBILITY:
Inclusion Criteria:

* Cases: Inaugural acute bronchiolitis in infant aged under 1 year; bronchiolitis is defined by rhinorrhea and/or cough, dyspnea, associated with clinical or radiological distension, wheezing or crackling or brake expiratory.
* Controls: Infant aged under 1 year with blood sample test performed for a non-infectious disease (preoperative assessment)

Exclusion Criteria:

* Cases: bronchopulmonary dysplasia, prematurity, cystic fibrosis, immunodeficiency, primary ciliary dyskinesia, congenital cardiopathy, use of corticotherapy the week between inclusion
* Controls: infectious documented disease, respiratory symptoms

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: infants aged under 1 year
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-10; Primary Completion 2016-05 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
KL-6 rate | At day 1

CONTACTS AND LOCATIONS:
Overall Officials: André LABBE, PU PH, Principal Investigator — CHU Estaing